CLINICAL TRIAL: NCT01161290
Title: A Randomized Controlled Trial Using Real-Time Interactive Audio/Visual Telehealth to Promote Self-care Management for United States Veterans With Chronic Obstructive Pulmonary Disease: a Pilot Study
Brief Title: Real-Time Telehealth to Promote Self-care Management for Chronic Obstructive Pulmonary Disease
Acronym: E-Breathe
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Breathe California, Los Angeles County (Other)
Responsible Party: Margaret Nield, Greater Los Angeles Healthcare System, West Los Angeles
Organization: VA Greater Los Angeles Healthcare System (U.S. Federal Agency)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: Nield005; BBRI 900.1553 (Other Grant/Funding Number: Breathe California, Los Angeles County)
Record Dates: First submitted 2010-07-12; First posted 2010-07-13 (Estimated); Last update posted 2010-07-13 (Estimated); Status verified 2010-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Telemedicine; Internet; Dyspnea; Self care; Breathing Exercises; Real-Time Systems
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: synchronous interactive audio/video telecommunication — 4 weekly synchronous interactive audio/video sessions on self-care management for dyspnea provided via the Internet and free downloadable software (Skype) on patients' home computer
  Other Names: Skype

SUMMARY:
HYPOTHESIS:The study purpose is to evaluate the effectiveness of a structured pursed-lips breathing (PLB) protocol taught via real-time interactive telecommunication with a home computer using the lnternet and Skype software in veterans with chronic obstructive pulmonary disease (COPD. The primary hypothesis is veterans with COPD and dyspnea on exertion who receive a PLB educational intervention taught via weekly interactive telecommunication over a 4-week period will have greater reduction of exertional dyspnea compared to those who receive the PLB educational intervention with no weekly interactive sessions.

RESEARCH PLAN: An experimental two- group design is used. All subjects receive a brief 5 - 10 minute one-on-one PLB educational session. Subjects are then randomized to either the intervention group or the control group. The intervention group receives 4 weekly interactive group sessions with the health educator (principal investigator)via computer. A free software program known as Skype allows synchronous video and audio interaction. The comparison group receives only the brief PLB educational session with no weekly follow-up.

RESULTS: At end of 4 weeks, the intervention group had significantly lower dyspnea intensity scores (group X time interaction F = 6.69, p = 0.02) and significantly higher social support scores (group x time interaction F = 4.34, p = 0.058).

CLINICAL SIGNIFICANCE: Skype is a viable means for providing patient education. A structured PLB protocol provides significant differences in exertional dyspnea over time. A structured PLB protocol plus Skype showed significant reduction in patients' sense of dyspnea intensity and increased social support scores.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of COPD, expiratory airflow limitation evidenced by forced expiratory volume 1 second/forced vital capacity percent (FEV1/FVC %) less than 70 and FEV1 % predicted less than 80 with no reversibility by inhaled bronchodilator, and self report of shortness of breath when walking as assessed with the modified Medical Research Council (MRC) chronic dyspnea questionnaire.

-

Exclusion Criteria:

Exacerbation of symptoms (dyspnea, increased sputum volume, and/or increased sputum purulence) within the past four weeks, hospital admission within the past four weeks, change in bronchodilator therapy within the past two weeks, unable to walk, unstable angina, unstable cardiac dysrhythmia, unstable congestive heart failure, and/or unstable neurosis or psychiatric disturbance.

-

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-09; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Dyspnea Intensity | End of 4 weeks and end of 12 weeks
  Dyspnea Intensity is measured with the Visual Analogue Scale. The scale is a 100-cm horizontal line with verbal anchors at either end. Interval level data are obtained by measuring from left to the point marked by the subject. The subjects mark the scale with a pencil in response to the question, "During the last 24 hours, how easy or how hard was it to get your breath?"

CONTACTS AND LOCATIONS:
Overall Officials: Margaret A Nield, PhD, Principal Investigator — Greater Los Angeles Healthcare System